CLINICAL TRIAL: NCT00963417
Title: TEXT-Bone: A Substudy of the TEXT Trial to Evaluate Serial Bone Markers for Bone Remodeling, Serial Growth Factors, and Bone Mineral Density
Brief Title: Study of Bone Mineral Density in Women With Breast Cancer Treated With Triptorelin and Tamoxifen or Exemestane on Protocol IBCSG 25-02
Acronym: TEXT-Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000637437; IBCSG-25A-02; BIG-25A-02; NABCI-IBCSG-25A-02
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triptorelin plus tamoxifen (Active Comparator): Determination of bone mineral density in patients randomized in TEXT-1 or TEXT-2 trials to receive triptorelin (GnRH analogue) for 5 years plus tamoxifen for 5 years.
  Interventions: Other: laboratory biomarker analysis; Procedure: dual x-ray absorptiometry
- Triptorelin plus exemestane (Experimental): Determination of bone mineral density in patients randomized in TEXT-1 or TEXT-2 trials to receive triptorelin (GnRH analogue) for 5 years plus exemestane for 5 years.
  Interventions: Other: laboratory biomarker analysis; Procedure: dual x-ray absorptiometry

INTERVENTIONS:
Other: laboratory biomarker analysis — Serial serum levels of several biomarkers will be analyzed at different time points, up to 72 months after randomization.
Procedure: dual x-ray absorptiometry — Serial bone mineral density measurements of the L1-L4 (postero-anterior, PA) region of the spine and hip by dual-energy X-ray absorptiometry (DEXA).

SUMMARY:
RATIONALE: Gathering information over time from bone density and laboratory tests of women with breast cancer treated with triptorelin and tamoxifen or exemestane may help the study of breast cancer in the future.

PURPOSE: This clinical trial is studying changes in bone mineral density in women with breast cancer treated with triptorelin and tamoxifen or exemestane on protocol IBC SG-25-02 (TEXT).

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate changes in bone mineral density (BMD) among premenopausal women randomized in protocol IBC SG-25202 (TEXT-2) to receive either: A) triptorelin (GnRH analogue) for 5 years plus tamoxifen for 5 years; or B) triptorelin (GnRH analogue) for 5 years plus the steroidal aromatase inhibitor exemestane for 5 years.
* Evaluate serial serum markers for bone remodeling (C-telopeptide, osteocalcin, bone-specific alkaline phosphatase) and investigate their correlation with BMD.
* Evaluate the relationship of genetic variants of CYP19A1, ERα, ERß, and IGF 1 with BMD.
* Evaluate serial serum growth factors (IGF-1 and IGFBP-3) and investigate whether their time course correlates with BMD.
* Explore the role of serum IGF-1 and IGFBP-3 as biomarkers of disease outcome (disease-free survival). (exploratory)

OUTLINE: Blood samples are collected at baseline and then periodically for 6 years. Serum markers of bone remodeling and serum growth factor levels are measured.

Bone mineral density in the L1-L4 (postero-anterior) region of the spine and femoral neck of the hip is measured by DEXA at baseline and then periodically for 6 years.

Any surplus serum is stored for use in unspecified future research.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient must be eligible and enrolled in the TEXT-2 trial prior to enrolling in TEXT-Bone
* Serial bone marrow density (BMD) measurements must be taken within the same institution
* Hormone receptor positive

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Premenopausal
* No bone fracture in the past 6 months that, in the investigator's judgement, could be related to bone fragility
* No clinical or biochemical malabsorption syndrome, known vitamin D deficiency, active hyper- or hypoparathyroidism, or Paget's disease
* No uncontrolled thyroid disease, Cushing disease, or other pituitary diseases
* No other bone disease (including osteomalacia or osteogenesis imperfecta)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 months since prior and no concurrent bisphosphonate therapy (or other bone therapies such as PTH or strontium)
* At least 6 months since prior glucocorticoid (> 5 mg prednisone or equivalent) for > 1 month
* At least 12 months since prior anticonvulsants

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-08-03 (Actual); Primary Completion 2011-03-11 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Serial serum levels of C-telopeptide, osteocalcin, and bone-specific alkaline phosphatase | 72 months after rnadomization to TEXT Study
Serial serum levels of IGF-1 and IGFBP-3 | 72 months after randomization to TEXT Study
Serial BMD measurements of the L1-L4 (postero-anterior, PA) region of the spine and hip by dual-energy X-ray absorptiometry (DEXA) | 72 months after randomization to TEXT Study

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Pagani, MD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni
Locations (13):
- Australia (5):
  - Royal Brisbane and Women's Hospital, Brisbane
  - Peter MacCallum Cancer Center, East Melbourne
  - Box Hill Hospital, Melbourne
  - Maroondah Hospital, Melbourne
  - Royal Perth Hospital, Perth
- Belgium (5):
  - Centre Hospitalier Regional de Huy, Huy
  - UZ Leuven, Leuven
  - C.H.U. Sart Tilman, Liège
  - CHR Citadelle, Liège
  - C.H.P.L.T. de Verviers, Verviers
- Switzerland (3):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No